CLINICAL TRIAL: NCT03622359
Title: Radiotracer Imaging of Skeletal Muscle Perfusion in Patients With Peripheral Artery Disease
Brief Title: Radiotracer-Based Perfusion Imaging of Patients With Peripheral Arterial Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Mitchel Stacy, Principal Investigator / Assistant Professor, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB18-00442
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Artery Disease; Diabetes Mellitus; Chronic Limb-Threatening Ischemia
Keywords: Radionuclide imaging; Perfusion imaging; Positron emission tomography; Single photon emission computed tomography
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPECT/CT perfusion imaging (Experimental): Patients with peripheral artery disease will have already been scheduled for clinically indicated revascularization procedures of the lower extremity and undergo SPECT/CT imaging as part of the research protocol.
  Interventions: Diagnostic Test: SPECT/CT perfusion imaging; Diagnostic Test: PET/CT perfusion imaging
- PET/CT perfusion imaging (Experimental): Patients with peripheral artery disease will have already been scheduled for clinically indicated revascularization procedures of the lower extremity and undergo PET/CT imaging as part of the research protocol.
  Interventions: Diagnostic Test: SPECT/CT perfusion imaging; Diagnostic Test: PET/CT perfusion imaging

INTERVENTIONS:
Diagnostic Test: SPECT/CT perfusion imaging — Subjects will receive a standard clinical dose of a radionuclide for perfusion imaging of the lower extremities before and after revascularization procedures.
Diagnostic Test: PET/CT perfusion imaging — Subjects will receive a standard clinical dose of a radionuclide for perfusion imaging of the lower extremities before and after revascularization procedures.

SUMMARY:
The aim of this clinical study is to 1) establish a healthy database for nuclear perfusion imaging of the lower extremities and 2) assess the prognostic value of radiotracer-based perfusion imaging for predicting clinical outcomes in patients with peripheral artery disease (PAD) who are undergoing lower extremity revascularization procedures. We hypothesize that radiotracer imaging of the lower extremities will provide a sensitive non-invasive imaging tool for quantifying regional abnormalities in skeletal muscle perfusion and evaluating responses to medical treatment.

DETAILED DESCRIPTION:
PAD patients (n=80) with peripheral artery disease (PAD) who are scheduled to undergo lower extremity revascularization procedures will be recruited. Patients will be screened using a standard medical history questionnaire and a physical activity questionnaire. Once their questionnaires are reviewed, individuals who meet inclusion criteria will proceed with standard PAD screening, which will include Ankle-Brachial Indices (ABIs) and Toe-Brachial Indices (TBIs) of both lower extremities. Patients will undergo SPECT/CT or PET/CT perfusion imaging prior to their revascularization procedure and 1-14 days following revascularization. Subjects will receive an intravenous injection of a standard clinical dose of radiotracer for both imaging sessions. A low-dose CT scan will be performed immediately after each SPECT and PET image acquisition for the purposes of attenuation correction and regional analysis of radiotracer uptake. Clinical outcomes will be evaluated for up to 12 months after the imaging study to assess the prognostic value of perfusion imaging for predicting subsequent outcomes. An additional subset of PAD patients (n=56) and healthy control subjects (n=56) will be enrolled to undergo the same imaging procedures to establish a healthy database for PET perfusion imaging measures.

ELIGIBILITY:
Inclusion Criteria for Patients with Peripheral Artery Disease:

1. At least 18 years of age
2. Evidence of significant obstructive disease for one or multiple lower extremity arteries, as identified by prior ABI, TBI, CT angiography, ultrasound, or MR imaging.

Exclusion Criteria for Patients with Peripheral Artery Disease:

1. Unable to give informed consent or follow-up
2. Pregnant or nursing
3. Under the age of 18
4. No history of peripheral artery disease

Inclusion Criteria for Healthy Control Subjects:

1. At least 18 years of age
2. No evidence or prior diagnosis of peripheral artery disease based on chart review and standard vascular screening.

Exclusion Criteria for Healthy Control Subjects:

1. Unable to give informed consent of follow-up
2. Pregnant or nursing
3. Under the age of 18
4. History of peripheral artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower extremity perfusion | 1-2 weeks
  The percent or absolute change in perfusion from baseline to post-revascularization will be evaluated.

SECONDARY OUTCOMES:
Wound healing | 1 year
  Rates of wound healing will be documented for 12 months following enrollment into the imaging study.
Limb salvage | 1 year
  Amputation rates will be documented for the 12 months following enrollment into the imaging study.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel R Stacy, Ph.D., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvelo JL, Papademetris X, Mena-Hurtado C, Jeon S, Sumpio BE, Sinusas AJ, Stacy MR. Radiotracer Imaging Allows for Noninvasive Detection and Quantification of Abnormalities in Angiosome Foot Perfusion in Diabetic Patients With Critical Limb Ischemia and Nonhealing Wounds. Circ Cardiovasc Imaging. 2018 May;11(5):e006932. doi: 10.1161/CIRCIMAGING.117.006932. PMID 29748311
- [Background] Chou TH, Atway SA, Bobbey AJ, Sarac TP, Go MR, Stacy MR. SPECT/CT Imaging: A Noninvasive Approach for Evaluating Serial Changes in Angiosome Foot Perfusion in Critical Limb Ischemia. Adv Wound Care (New Rochelle). 2020 Mar 1;9(3):103-110. doi: 10.1089/wound.2018.0924. Epub 2020 Jan 24. PMID 31993252
- [Background] Chou TH, Stacy MR. Clinical Applications for Radiotracer Imaging of Lower Extremity Peripheral Arterial Disease and Critical Limb Ischemia. Mol Imaging Biol. 2020 Apr;22(2):245-255. doi: 10.1007/s11307-019-01425-3. PMID 31482412
- [Background] Chou TH, Tram NK, Eisert SN, Bobbey AJ, Atway SA, Go MR, Stacy MR. Dual assessment of abnormal microvascular foot perfusion and lower extremity calcium burden in a patient with critical limb ischemia using hybrid SPECT/CT imaging. Vasc Med. 2021 Apr;26(2):225-227. doi: 10.1177/1358863X20964563. Epub 2020 Oct 30. No abstract available. PMID 33126838
- [Background] Chou TH, Alvelo JL, Janse S, Papademetris X, Sumpio BE, Mena-Hurtado C, Sinusas AJ, Stacy MR. Prognostic Value of Radiotracer-Based Perfusion Imaging in Critical Limb Ischemia Patients Undergoing Lower Extremity Revascularization. JACC Cardiovasc Imaging. 2021 Aug;14(8):1614-1624. doi: 10.1016/j.jcmg.2020.09.033. Epub 2020 Nov 18. PMID 33221224
- [Background] Tram NK, Chou TH, Patel S, Ettefagh LN, Go MR, Atway SA, Stacy MR. Novel Application of 18F-NaF PET/CT Imaging for Evaluation of Active Bone Remodeling in Diabetic Patients With Charcot Neuropathy: A Proof-of-Concept Report. Front Med (Lausanne). 2022 Feb 18;9:795925. doi: 10.3389/fmed.2022.795925. eCollection 2022. PMID 35252240
- [Background] Stacy MR. Molecular Imaging of Lower Extremity Peripheral Arterial Disease: An Emerging Field in Nuclear Medicine. Front Med (Lausanne). 2022 Jan 12;8:793975. doi: 10.3389/fmed.2021.793975. eCollection 2021. PMID 35096884
- [Background] Rimmerman ET, Musini KN, Chou TH, Wynveen MK, Patel SA, Beall M, Bobbey AJ, Atway SA, Go MR, Stacy MR. Vessel-by-Vessel Computed Tomography Calcium Scoring of the Foot in Peripheral Artery Disease: Association with Patient-Level Factors. Adv Wound Care (New Rochelle). 2023 Nov;12(11):603-610. doi: 10.1089/wound.2022.0151. Epub 2023 Feb 7. PMID 36601736
- [Background] Chou TH, Rimmerman ET, Patel S, Wynveen MK, Eisert SN, Musini KN, Janse SA, Bobbey AJ, Sarac TP, Atway SA, Go MR, Stacy MR. Vessel-by-vessel analysis of lower extremity 18F-NaF PET/CT imaging quantifies diabetes- and chronic kidney disease-induced active microcalcification in patients with peripheral arterial disease. EJNMMI Res. 2023 Jan 17;13(1):3. doi: 10.1186/s13550-023-00951-0. PMID 36648583
- [Background] Chou TH, Wynveen MK, Rimmerman ET, Patel S, Go MR, Stacy MR. Detection of multivessel calcific disease progression in a patient with chronic limb-threatening ischemia using fluorine-18 sodium fluoride positron emission tomography imaging. J Vasc Surg Cases Innov Tech. 2023 Mar 4;9(2):101137. doi: 10.1016/j.jvscit.2023.101137. eCollection 2023 Jun. PMID 37139350
- [Background] Chou TH, Nabavinia M, Tram NK, Rimmerman ET, Patel S, Musini KN, Eisert SN, Wolfe T, Wynveen MK, Matsuzaki Y, Kitsuka T, Iwaki R, Janse SA, Bobbey AJ, Breuer CK, Goodchild L, Malbrue R, Shinoka T, Atway SA, Go MR, Stacy MR. Quantification of Skeletal Muscle Perfusion in Peripheral Artery Disease Using 18F-Sodium Fluoride Positron Emission Tomography Imaging. J Am Heart Assoc. 2024 Feb 20;13(4):e031823. doi: 10.1161/JAHA.123.031823. Epub 2024 Feb 14. PMID 38353265